CLINICAL TRIAL: NCT01659021
Title: A Phase 3, Randomized, Controlled Study Evaluating the Efficacy and Safety of Idelalisib (GS-1101) in Combination With Ofatumumab for Previously Treated Chronic Lymphocytic Leukemia
Brief Title: Efficacy and Safety of Idelalisib in Combination With Ofatumumab for Previously Treated Chronic Lymphocytic Leukemia
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-312-0119; 2012-001236-65 (EudraCT Number)
Record Dates: First submitted 2012-08-03; First posted 2012-08-07 (Estimated); Results first posted 2017-03-31 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: CLL; Chronic Lymphocytic Leukemia; GS-1101; CAL-101; Ofatumumab
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — idelalisib; ofatumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Idelalisib+ofatumumab (Experimental): Randomized Initial Therapy (24 weeks): Idelalisib + ofatumumab for a total of 12 infusions (300 mg on Day 1, followed by 1000 mg weekly for 7 weeks, and then 1000 mg every 4 weeks for 4 doses)
  Continuing Therapy/Observation: Idelalisib 150 mg tablets twice daily until the earliest of participant withdrawal from study, definitive progression of CLL, intolerable idelalisib-related toxicity, pregnancy or initiation of breast feeding, substantial noncompliance with study procedures, or study discontinuation.
  Long-Term Follow-up: Participants were followed for up to 5 years. Information on medical status, anti-tumor treatments, secondary malignancies, and survival status were collected annually during a routine clinic visit or other contact, such as telephone.
  Interventions: Drug: Idelalisib; Drug: Ofatumumab
- Ofatumumab (Active Comparator): Randomized Initial Therapy (24 weeks): Ofatumumab for a total of 12 infusions (300 mg on Day 1, followed by 2000 mg weekly for 7 weeks, and then 2000 mg every 4 weeks for 4 doses)
  Continuing Therapy/Observation: Observation until the earliest of participant withdrawal from study, definitive progression of CLL, intolerable idelalisib-related toxicity, pregnancy or initiation of breast feeding, substantial noncompliance with study procedures, or study discontinuation.
  Long-Term Follow-up: Participants were followed for up to 5 years. Information on medical status, anti-tumor treatments, secondary malignancies, and survival status were collected annually during a routine clinic visit or other contact, such as telephone.
  Interventions: Drug: Ofatumumab

INTERVENTIONS:
Drug: Idelalisib — 150 mg tablets administered orally twice daily
  Other Names: Zydelig®; GS-1101; CAL-101
  Arms: Idelalisib+ofatumumab
Drug: Ofatumumab — Administered intravenously
  Other Names: Arzerra®

SUMMARY:
The primary objective of this study is to evaluate the effect of the addition of idelalisib to ofatumumab on progression-free survival (PFS) in participants with previously treated chronic lymphocytic leukemia (CLL).

ELIGIBILITY:
Key Inclusion Criteria:

* Adults with previously treated recurrent CLL who have measurable lymphadenopathy
* Require therapy for CLL
* Have experienced CLL progression < 24 months since the completion of the last prior therapy
* Have disease that is not refractory to ofatumumab

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 261 (Actual)
Dates: Start 2012-12-04 (Actual); Primary Completion 2018-08-15 (Actual); Study Completion 2018-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (79):
- United States (24):
  - City of Hope, Duarte, California
  - California Cancer Associates for Research and Excellence (CCARE), Fresno, California
  - Kaiser Permanente, San Diego, California
  - Coastal Integrative Cancer Care, San Luis Obispo, California
  - Stanford University Medical Center, Stanford, California
  - Kaiser Permanente Vallejo Medical Center, Vallejo, California
  - Kaiser Permanente of Colorado, Denver, Colorado
  - Saint Mary's Regional Cancer Center, Grand Junction, Colorado
  - Cancer Specialists of North Florida, Jacksonville, Florida
  - Georgia Regents University, Augusta, Georgia
  - Montgomery Cancer Center, Mount Sterling, Kentucky
  - Center for Cancer and Blood Disorders, PC, Bethesda, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Washington University Medical Center, St Louis, Missouri
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Weill Cornell Medical Center, New York, New York
  - Oncology Hematology Care, Inc., Cincinnati, Ohio
  - The Ohio State University Medical Center, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Upstate Oncology Associates, Greenville, South Carolina
  - Tennessee Oncology, PLLC, Chattanooga, Tennessee
  - Tenessee Oncology, PLLC, Nashville, Tennessee
  - Utah Cancer Specialists, Salt Lake City, Utah
  - Northwest Medical Specialties, Tacoma, Washington
- Australia (9):
  - Saint George and Sutherland Hospitals, Kogarah, New South Wales
  - Prince of Wales Hospital, Randwick, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Haematology and Oncology Clinics of Australia at Mater, Milton, Queensland
  - Ashford Cancer Centre Research, Ashford, South Australia
  - Box Hill Hospital, Box Hill, Victoria
  - Frankston Hospital, Melbourne, Victoria
  - Queen Elizabeth Hospital, Woodville
- Belgium (4):
  - Ziekenhuis Netwerk Antwerpen, Antwerp
  - Cliniques Universitaires Saint Luc, Brussels
  - Universitair Ziekenhuis Gent, Ghent
  - Universitaire Ziekenhuis Gasthuisberg, Leuven
- Canada (8):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - Cancer Care Manitoba, Winnipeg, Manitoba
  - Hopital Regional De Sudbury Regional Hospital (HRSRH) - Regional Cancer Program (RCP), Greater Sudbury, Ontario
  - Centre Hospitalier Universitaire de Montréal, Montreal, Quebec
  - Centre Hospitalier Regional de Rimouski, Rimouski, Quebec
  - Saskatchewan Cancer Agency, Regina, Saskatchewan
  - Cancer Care Manitoba, Winnipeg
- Denmark (2):
  - Aalborg Hospital, Aalborg
  - Aarhus University Hospital, Aarhus
- France (7):
  - Center Hospitalier Universitaire de Bordeaux, Pessac, Aquitaine
  - Centre Hospitalier de Perpignan, Perpignan, Languedoc-Roussillon
  - Centre Hospitalier Universitaire Nancy, Vandœuvre-lès-Nancy, Limousin, Lorraine
  - Centre Hospitalier Universitaire Purpan, Toulouse, Midi-pyrenees
  - CHRU Clermont- Ferrand CHU Estaing, Auvergne
  - Centre Hospitalier Universitaire Hôpital Avicenne, Ile-de-france
  - Hôpital Saint Louis, Paris, Île-de-France Region
- Ireland (2):
  - University College Cork, Cork
  - Saint James's Hospital, Dublin
- Poland (6):
  - Collegium Medicum Uniwersytetu Jagiellonskiego w K, Krakow, Lesser Poland Voivodeship
  - Wojewódzki Szpital Specjalistyczny im. Janusza Kor, Słupsk, Pomeranian Voivodeship
  - Szpital Specjalistyczny w Brzozowie, Brzozów
  - Wojewódzki Szpital Specjalistyczny im. Mikolaja Kopernika w Lodzi, Lódz
  - Centralny Szpital Kliniczny MSW, Warsaw
  - Samodzielny Publiczny Szpital Kliniczny N1 Klinika, Wroclaw
- Spain (6):
  - Hospital Clínic i Provincial, Barcelona
  - Hospital Vall d´Hebrón, Barcelona
  - Hospital Universitario La Princesa, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Puerta de Hierro Majadahonda, Madrid
  - Hospital Morales Meseguer, Murcia
- Sweden (3):
  - Sunderby Sjukhus, Luleå
  - Karolinska University Hospital Solna, Stockholm
  - Karolinska University Hospital Huddinge, Stockholm
- United Kingdom (8):
  - Birmingham Heartlands Hospital, Birmingham, England
  - Darent Valley Hospital, Dartford, England
  - Royal Surrey County Hospital NHS Trust, Guildford, England
  - Haematology and Transplant Unit, Manchester, England
  - Norfolk and Norwich University Hospital, Norwich, Norfolk
  - Saint James's University Hospital, Leeds
  - University College London, London
  - Department of Haematology, Cancer and Haematology Centre, Churchill Hospital (Oxford University Hospitals), Oxford

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at http://www.gilead.com/research/disclosure-and-transparency.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: http://www.gilead.com/research/disclosure-and-transparency

REFERENCES:
- [Result] Jones JA, Robak T, Brown JR, Awan FT, Badoux X, Coutre S, Loscertales J, Taylor K, Vandenberghe E, Wach M, Wagner-Johnston N, Ysebaert L, Dreiling L, Dubowy R, Xing G, Flinn IW, Owen C. Efficacy and safety of idelalisib in combination with ofatumumab for previously treated chronic lymphocytic leukaemia: an open-label, randomised phase 3 trial. Lancet Haematol. 2017 Mar;4(3):e114-e126. doi: 10.1016/S2352-3026(17)30019-4. PMID 28257752
- [Result] Jones J, Robak T, Wach M, Brown JR, Menter AR, Vandenberghe E, et al. Updated results of a phase 3 randomized, controlled study of idelalisib in combination with ofatumumab for previously treated chronic lymphocytic leukemia (CLL) [Poster 7515]. American Society of Clinical Oncology (ASCO) 52nd Annual Meeting; 2016 02 - 06 June; Chicago, IL.
- [Result] Jones JA, Wach M, Robak T, Brown JR, Menter AR, Vanderberghe E, et al. Results of a Phase 3 Randomized, Controlled Study Evaluating the Efficacy and Safety of Idelalisib (IDELA) in Combination with Ofatumumab (OFA) for Previously Treated Chronic Lymphocytic Leukemia (CLL) [Poster 7023]. American Society of Clinical Oncology (ASCO) 51st Annual Meeting; 2015 29 May - 02 June; Chicago, IL.
- [Result] Robak T, Jones J, Wach M, Brown JR, Menter AR, Vandenberghe E, et al. Updated results of a phase 3 randomized, controlled study of idelalisib in combination with ofatumumab for previously treated chronic lymphocytic leukemia (CLL) [Poster 213]. 21st Congress of the European Hematology Association (EHA); 2015 09-12 June; Copenhagen, Denmark.
- [Result] Robak T, Wach M, Jones J, Owen C, Brown J, Menter A, et al. Results Of A Phase 3 Randomized Controlled Study Evaluating The Efficacy And Safety Of Idelalisib (Idela) In Combination With Ofatumumab (Ofa) For Previously Treated Chronic Lymphocytic Leukemia (CLL) [Poster LB598]. 20th Congress of the European Hematology Association (EHA); 2015 11-14 June; Vienna, Austria.
- [Result] Flinn I, Kimby E, Cotter FE, Giles FJ, Janssens A, Pulczynski EJ, et al. A Phase 3, Randomized, Controlled Study Evaluating the Efficacy and Safety of Idelalisib (GS-1101) in Combination with Ofatumumab for Previously Treated Chronic Lymphocytic Leukemia (CLL) [Poster TPS7131]. American Society of Clinical Oncology (ASCO); 2013 May 31-June 4; Chicago, IL.
- [Derived] Gordon MJ, Huang J, Chan RJ, Bhargava P, Danilov AV. Medical comorbidities in patients with chronic lymphocytic leukaemia treated with idelalisib: analysis of two large randomised clinical trials. Br J Haematol. 2021 Feb;192(4):720-728. doi: 10.1111/bjh.16879. Epub 2020 Jun 29. PMID 32599655

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in North America, Europe, and Australia. The first participant was screened on 04 December 2012. The last study visit occurred on 15 August 2018.
Pre-assignment Details: 310 participants were screened.
Groups:
- Idelalisib+Ofatumumab: Randomized Initial Therapy (24 weeks): Idelalisib 150 mg tablets twice daily + ofatumumab for a total of 12 infusions (300 mg on Day 1, followed by 1000 mg weekly for 7 weeks, and then 1000 mg every 4 weeks for 4 doses)
  Continuing Therapy/Observation: Idelalisib 150 mg tablets twice daily until the earliest of subject withdrawal from study, definitive progression of chronic lymphocytic leukemia (CLL), intolerable idelalisib-related toxicity, pregnancy or initiation of breast feeding, substantial noncompliance with study procedures, or study discontinuation
  Long-Term Follow-up: Participants were followed for up to 5 years. Information on medical status, anti-tumor treatments, secondary malignancies, and survival status were collected annually during a routine clinic visit or other contact, such as telephone.
- Ofatumumab: Randomized Initial Therapy (24 weeks): Ofatumumab for a total of 12 infusions (300 mg on Day 1, followed by 2000 mg weekly for 7 weeks, and then 2000 mg every 4 weeks for 4 doses)
  Continuing Therapy/Observation: Observation until the earliest of subject withdrawal from study, definitive progression of CLL, intolerable idelalisib-related toxicity, pregnancy or initiation of breast feeding, substantial noncompliance with study procedures, or study discontinuation
  Long-Term Follow-up: Participants were followed for up to 5 years. Information on medical status, anti-tumor treatments, secondary malignancies, and survival status were collected annually during a routine clinic visit or other contact, such as telephone.
Period: Main Study
Arm/Group | Idelalisib+Ofatumumab | Ofatumumab
Started | 174 | 87
Randomized and Treated | 173 | 86
Completed (Study completion was defined as disease progression or death.) | 100 | 50
Not Completed | 74 | 37
Not completed — Adverse Event | 2 | 3
Not completed — Lost to Follow-up | 1 | 0
Not completed — Unknown Reasons | 2 | 1
Not completed — Physician Decision | 34 | 16
Not completed — Withdrawal by Subject | 19 | 16
Not completed — Study Terminated by Sponsor | 16 | 1
Period: Long-Term Follow Up
Arm/Group | Idelalisib+Ofatumumab | Ofatumumab
Started | 138 (Participants did not have to complete the main study to enter the Long-Term Follow Up period.) | 69 (Participants did not have to complete the main study to enter the Long-Term Follow Up period.)
Completed | 133 | 65
Not Completed | 5 | 4
Not completed — Lost to Follow-up | 3 | 3
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) Analysis Set included participants who were randomized in the study regardless of whether they received any study drug(s), or received a different regimen from that to which they were randomized. Treatment assignment was designated according to randomization.
Groups:
- Idelalisib+Ofatumumab: Randomized Initial Therapy (24 weeks): Idelalisib 150 mg tablets twice daily + ofatumumab for a total of 12 infusions (300 mg on Day 1, followed by 1000 mg weekly for 7 weeks, and then 1000 mg every 4 weeks for 4 doses)
  Continuing Therapy/Observation: Idelalisib 150 mg tablets twice daily until the earliest of subject withdrawal from study, definitive progression of CLL, intolerable idelalisib-related toxicity, pregnancy or initiation of breast feeding, substantial noncompliance with study procedures, or study discontinuation
- Ofatumumab: Randomized Initial Therapy (24 weeks): Ofatumumab for a total of 12 infusions (300 mg on Day 1, followed by 2000 mg weekly for 7 weeks, and then 2000 mg every 4 weeks for 4 doses)
  Continuing Therapy/Observation: Observation until the earliest of subject withdrawal from study, definitive progression of CLL, intolerable idelalisib-related toxicity, pregnancy or initiation of breast feeding, substantial noncompliance with study procedures, or study discontinuation
- Total: Total of all reporting groups
Arm/Group | Idelalisib+Ofatumumab | Ofatumumab | Total
Number analyzed (Participants) | 174 | 87 | 261
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (9.0) | 67 (9.7) | 67 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 25 | 75
  Male | 124 | 62 | 186
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 3 | 10
  Not Hispanic or Latino | 141 | 74 | 215
  Unknown or Not Reported | 26 | 10 | 36
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 149 | 71 | 220
  Black or African American | 0 | 4 | 4
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Asian | 2 | 0 | 2
  Other | 2 | 3 | 5
  Not Permitted | 20 | 9 | 29
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 13 | 9 | 22
  Sweden | 4 | 2 | 6
  Belgium | 5 | 1 | 6
  United States | 64 | 29 | 93
  Ireland | 7 | 4 | 11
  Denmark | 4 | 0 | 4
  Poland | 27 | 9 | 36
  United Kingdom | 11 | 6 | 17
  Australia | 16 | 13 | 29
  France | 15 | 9 | 24
  Spain | 8 | 5 | 13
Time Since Diagnosis [Mean (Standard Deviation); unit: months] — Population: Only participants who were randomized and treated are included.
  months
    number analyzed (Participants) | 173 | 86 | 259
    (all) | 101.0 (60.21) | 94.3 (52.51) | 98.8 (57.75)
17p deletion and/or TP53 mutation [Count of Participants; unit: Participants]
  Either | 70 | 33 | 103
  Neither | 104 | 54 | 158
Immunoglobulin heavy chain variable region (IGHV) mutation status [Count of Participants; unit: Participants]
  Mutated | 37 | 19 | 56
  Unmutated | 137 | 68 | 205
Disease Status [Count of Participants; unit: Participants] — Refractory: CLL progression < 6 months from completion of prior therapy; Relapsed: CLL progression ≥ 6 months from completion of prior therapy.
  Participants
    Refractory | 82 | 47 | 129
    Relapsed | 92 | 40 | 132

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival
Description: Progression-free survival (PFS) was defined as the interval from randomization to the earlier of the first documentation of definitive disease progression or death from any cause. Definitive disease progression was CLL progression based on standard criteria (other than lymphocytosis alone) as defined by the 2008 update of the International Workshop on CLL guidelines, ie, appearance of any new lesion; increase by ≥ 50% in the sum of the products of the perpendicular diameters of measured lymph nodes (SPD); new or ≥ 50% enlargement of liver or spleen; transformation to a more aggressive histology (eg, Richter's or prolymphocytic transformation); reduction in the number of blood cells (cytopenia) attributable to CLL. PFS was analyzed using Kaplan-Meier (KM) estimates.
Time Frame: Randomization to End of Study (up to 60 months)
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Idelalisib+Ofatumumab | Ofatumumab
Number analyzed (Participants) | 174 | 87
months | 16.6 [13.7 to 19.6] | 8.0 [5.7 to 8.4]
Statistical Analysis 1: Comparison: Idelalisib+Ofatumumab vs Ofatumumab; Test type: Superiority; p < 0.0001, Log Rank — P-value is from stratified log-rank test, adjusted for randomization stratification factors (17p deletion/TP53 mutation, immunoglobulin heavy chain variable region (IGHV) mutation, and disease status); Hazard Ratio (HR) = 0.26, 95% CI 2-sided [0.18 to 0.37] — Hazard Ratio and 95% confidence intervals (CI) are from the proportional hazard model, adjusted for randomization stratification factors

2. Secondary Outcome: Overall Response Rate
Description: Overall response rate was defined as the percentage of participants who achieved a best overall response of complete response or partial response.
  * Complete response was defined as no lymphadenopathy, hepatomegaly, splenomegaly; normal complete blood count; confirmed by bone marrow aspirate & biopsy.
  * Partial response was defined as >1 of the following criteria: a 50% decrease in peripheral blood lymphocytes, lymphadenopathy, liver size, spleen size; plus ≥ 1 of the following: ≥ 1500/μL absolute neutrophil count, > 100000/μL platelets, > 11.0 g/dL hemoglobin or 50% improvement for either of these parameters without transfusions or growth factors. Overall response rate was analyzed using KM estimates.
Time Frame: Randomization to End of Study (up to 60 months)
Population: Participants in the ITT Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Idelalisib+Ofatumumab | Ofatumumab
Number analyzed (Participants) | 174 | 87
percentage of participants | 75.3 [68.2 to 81.5] | 17.2 [10.0 to 26.8]
Statistical Analysis 1: Comparison: Idelalisib+Ofatumumab vs Ofatumumab; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was calculated from the Cochran-Mantel-Haenszel (CMH) Chi-square test stratified by stratification factors; Odds Ratio (OR) = 16.85, 95% CI 2-sided [8.17 to 34.76] — Odds ratio and 95% CIs were calculated from the CMH Chi-square test stratified by stratification factors

3. Secondary Outcome: Lymph Node Response Rate
Description: Lymph node response rate was defined as the proportion of participants who achieved a ≥ 50% decrease from baseline in the sum of the products of the greatest perpendicular diameters (SPD) of index lymph nodes.
Time Frame: Randomization to End of Study (up to 60 months)
Population: Participants in the ITT Analysis Set with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Idelalisib+Ofatumumab | Ofatumumab
Number analyzed (Participants) | 164 | 81
percentage of participants | 92.7 [87.6 to 96.2] | 4.9 [1.4 to 12.2]
Statistical Analysis 1: Comparison: Idelalisib+Ofatumumab vs Ofatumumab; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was calculated from the CMH Chi-square test stratified by stratification factors; Odds Ratio (OR) = 483.16, 95% CI 2-sided [94.63 to 2467.02] — Odds ratio and 95% CIs were calculated from the CMH Chi-square test stratified by stratification factors

4. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the interval from randomization to death from any cause. Overall survival was analyzed using KM estimates.
Time Frame: Randomization to Last Long-Term Follow-Up Visit (up to maximum of 5 years)
Population: Participants in the ITT Analysis Set were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Idelalisib+Ofatumumab: Randomized Initial Therapy (24 weeks): Idelalisib 150 mg tablets twice daily + ofatumumab for a total of 12 infusions (300 mg on Day 1, followed by 1000 mg weekly for 7 weeks, and then 1000 mg every 4 weeks for 4 doses)
  Continuing Therapy/Observation: Idelalisib 150 mg tablets twice daily until the earliest of subject withdrawal from study, definitive progression of CLL, intolerable idelalisib-related toxicity, pregnancy or initiation of breast feeding, substantial noncompliance with study procedures, or study discontinuation
  Long-Term Follow-up: Participants were followed for up to 5 years. Information on medical status, anti-tumor treatments, secondary malignancies, and survival status were collected annually during a routine clinic visit or other contact, such as telephone.
Arm/Group | Idelalisib+Ofatumumab | Ofatumumab
Number analyzed (Participants) | 174 | 87
months | 45.2 [34.1 to NA] — NA = Too few events to estimate the upper limit of the confidence interval. | 39 [23.0 to NA] — NA = Too few events to estimate the upper limit of the confidence interval.
Statistical Analysis 1: Comparison: Idelalisib+Ofatumumab vs Ofatumumab; Test type: Superiority; p = 0.247, Log Rank — P-value is from stratified log-rank test, adjusted for randomization stratification factors (17p deletion/TP53 mutation, IGHV mutation, and disease status); Hazard Ratio (HR) = 0.79, 95% CI 2-sided [0.54 to 1.15]

5. Secondary Outcome: Progression-Free Survival in Subgroup of Participants With Chromosome 17p Deletion and/or TP53 Mutation
Description: Progression-free survival in subgroup of participants with chromosome 17p deletion and/or TP53 mutation was analyzed using KM estimates.
Time Frame: Randomization to End of Study (up to 60 months)
Population: Participants in the ITT Analysis Set with chromosome 17p deletion and/or TP53 mutation were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Idelalisib+Ofatumumab: Randomized Initial Therapy (24 weeks): Idelalisib 150 mg tablets twice daily + ofatumumab for a total of 12 infusions (300 mg on Day 1, followed by 1000 mg weekly for 7 weeks, and then 1000 mg every 4 weeks for 4 doses)
  Continuing Therapy/Observation: Idelalisib 150 mg tablets twice daily until the earliest of subject withdrawal from study, definitive progression of CLL, intolerable idelalisib-related toxicity, pregnancy or initiation of breast feeding, substantial noncompliance with study procedures, or study discontinuation
  Participants in this group had 17p deletion and/or TP53 mutation.
- Ofatumumab: Randomized Initial Therapy (24 weeks): Ofatumumab for a total of 12 infusions (300 mg on Day 1, followed by 2000 mg weekly for 7 weeks, and then 2000 mg every 4 weeks for 4 doses)
  Continuing Therapy/Observation: Observation until the earliest of subject withdrawal from study, definitive progression of CLL, intolerable idelalisib-related toxicity, pregnancy or initiation of breast feeding, substantial noncompliance with study procedures, or study discontinuation
  Participants in this group had 17p deletion and/or TP53 mutation.
Arm/Group | Idelalisib+Ofatumumab | Ofatumumab
Number analyzed (Participants) | 70 | 33
months | 16.2 [11.1 to 19.1] | 5.8 [4.5 to 8.4]
Statistical Analysis 1: Comparison: Idelalisib+Ofatumumab vs Ofatumumab; Test type: Other; Hazard Ratio (HR) = 0.30, 95% CI 2-sided [0.17 to 0.51] — Hazard ratio and 95% CIs were calculated using the Cox proportional hazards model without any adjustments

6. Secondary Outcome: Complete Response Rate
Description: Complete response rate was defined as the percentage of participants who achieve a complete response and maintain their response for at least 8 weeks (with a 1-week window).
Time Frame: Randomization to End of Study (up to 60 months)
Population: Participants in the ITT Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Idelalisib+Ofatumumab | Ofatumumab
Number analyzed (Participants) | 174 | 87
percentage of participants | 1.1 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events: Start of Treatment to End of Treatment (up to 60 months) plus 30 days; All-Cause Mortality: Baseline to Last Long-Term Follow-Up Visit (up to maximum of 5 years)
Description: All-Cause Mortality was assessed in all randomized participants. All other adverse events were assessed in the Safety Analysis Set (participants who received ≥ 1 dose of study treatment, with treatment assignments designated according to the actual treatment received).
Arm/Group | Idelalisib+Ofatumumab | Ofatumumab
All-Cause Mortality (participants affected / at risk) | 87/174 | 40/87
Serious Adverse Events (participants affected / at risk) | 136/173 | 36/86
Other Adverse Events (participants affected / at risk) | 167/173 | 79/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Idelalisib+Ofatumumab (N=173) | Ofatumumab (N=86)
Anaemia (Blood and lymphatic system disorders) | 8 | 2
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 19 | 3
Granulocytopenia (Blood and lymphatic system disorders) | 2 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 13 | 2
Pancytopenia (Blood and lymphatic system disorders) | 2 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 2
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 2 | 0
Aortic valve disease (Cardiac disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 3 | 2
Bradycardia (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Cardiogenic shock (Cardiac disorders) | 2 | 0
Myocardial infarction (Cardiac disorders) | 2 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 0 | 1
Right ventricular failure (Cardiac disorders) | 1 | 0
External ear inflammation (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 7 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Abdominal wall haematoma (Gastrointestinal disorders) | 1 | 0
Anal fistula (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 13 | 0
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 23 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 1 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 0
Stomatitis (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 3 | 0
Asthenia (General disorders) | 2 | 1
Chest pain (General disorders) | 2 | 0
Death (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 1 | 0
Generalised oedema (General disorders) | 0 | 1
Impaired self-care (General disorders) | 1 | 0
Influenza like illness (General disorders) | 1 | 0
Pyrexia (General disorders) | 23 | 1
Strangulated hernia (General disorders) | 1 | 0
Systemic inflammatory response syndrome (General disorders) | 1 | 0
Bile duct obstruction (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 2 | 0
Anaphylactic shock (Immune system disorders) | 0 | 1
Abscess (Infections and infestations) | 0 | 1
Aspergillus infection (Infections and infestations) | 1 | 0
Atypical pneumonia (Infections and infestations) | 2 | 0
Bacteraemia (Infections and infestations) | 2 | 0
Bacterial sepsis (Infections and infestations) | 1 | 0
Biliary sepsis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 4 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 1 | 0
Candida infection (Infections and infestations) | 1 | 0
Candida pneumonia (Infections and infestations) | 0 | 1
Candida sepsis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 2 | 0
Chronic sinusitis (Infections and infestations) | 1 | 0
Cytomegalovirus colitis (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 0 | 1
Escherichia bacteraemia (Infections and infestations) | 0 | 1
Escherichia sepsis (Infections and infestations) | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 1
Folliculitis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Gastroenteritis salmonella (Infections and infestations) | 1 | 0
Genital herpes (Infections and infestations) | 1 | 0
H1N1 influenza (Infections and infestations) | 0 | 1
Herpes simplex (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Herpes zoster disseminated (Infections and infestations) | 1 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Listeria sepsis (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 7 | 2
Lung infection (Infections and infestations) | 4 | 0
Neutropenic sepsis (Infections and infestations) | 4 | 2
Pneumocystis jirovecii infection (Infections and infestations) | 1 | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 8 | 0
Pneumonia (Infections and infestations) | 27 | 9
Progressive multifocal leukoencephalopathy (Infections and infestations) | 0 | 2
Pseudomonal bacteraemia (Infections and infestations) | 2 | 0
Pseudomonal sepsis (Infections and infestations) | 1 | 0
Pseudomonas infection (Infections and infestations) | 0 | 1
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 3 | 2
Respiratory tract infection bacterial (Infections and infestations) | 1 | 0
Rhinovirus infection (Infections and infestations) | 1 | 0
Salmonellosis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 11 | 1
Septic shock (Infections and infestations) | 5 | 1
Sinusitis (Infections and infestations) | 2 | 0
Skin infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 7 | 0
Urosepsis (Infections and infestations) | 1 | 0
Varicella (Infections and infestations) | 0 | 1
Vascular device infection (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 1 | 0
Viral sepsis (Infections and infestations) | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 3 | 0
Overdose (Injury, poisoning and procedural complications) | 2 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
C-reactive protein increased (Investigations) | 1 | 0
Lymphocyte count decreased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 6 | 0
Platelet count decreased (Investigations) | 1 | 0
Transaminases increased (Investigations) | 1 | 0
Troponin increased (Investigations) | 0 | 1
Weight decreased (Investigations) | 1 | 1
White blood cell count decreased (Investigations) | 1 | 0
Cachexia (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 6 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 3 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 3 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 0
Pseudohyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Central nervous system leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Mycosis fungoides (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Aphasia (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Embolic stroke (Nervous system disorders) | 1 | 0
Facial paralysis (Nervous system disorders) | 1 | 0
Hemiparesis (Nervous system disorders) | 2 | 0
Hypotonia (Nervous system disorders) | 1 | 0
Locked-in syndrome (Nervous system disorders) | 1 | 0
Peroneal nerve palsy (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 2 | 0
Device occlusion (Product Issues) | 1 | 0
Bipolar I disorder (Psychiatric disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 0
Mania (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 5 | 0
Chronic kidney disease (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 2 | 0
Renal failure (Renal and urinary disorders) | 3 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Lower respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 7 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 6 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Haematoma (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 7 | 1
Peripheral artery aneurysm (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Idelalisib+Ofatumumab (N=173) | Ofatumumab (N=86)
Anaemia (Blood and lymphatic system disorders) | 38 | 7
Neutropenia (Blood and lymphatic system disorders) | 57 | 14
Thrombocytopenia (Blood and lymphatic system disorders) | 25 | 5
Tachycardia (Cardiac disorders) | 10 | 2
Abdominal pain (Gastrointestinal disorders) | 28 | 5
Abdominal pain upper (Gastrointestinal disorders) | 15 | 4
Colitis (Gastrointestinal disorders) | 17 | 0
Constipation (Gastrointestinal disorders) | 39 | 13
Diarrhoea (Gastrointestinal disorders) | 96 | 21
Dyspepsia (Gastrointestinal disorders) | 13 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 15 | 3
Nausea (Gastrointestinal disorders) | 62 | 23
Stomatitis (Gastrointestinal disorders) | 9 | 0
Vomiting (Gastrointestinal disorders) | 29 | 12
Asthenia (General disorders) | 27 | 9
Chest pain (General disorders) | 9 | 2
Chills (General disorders) | 27 | 13
Fatigue (General disorders) | 60 | 24
Influenza like illness (General disorders) | 14 | 1
Malaise (General disorders) | 10 | 1
Oedema peripheral (General disorders) | 35 | 9
Pain (General disorders) | 13 | 2
Peripheral swelling (General disorders) | 12 | 1
Pyrexia (General disorders) | 55 | 19
Hypogammaglobulinaemia (Immune system disorders) | 11 | 3
Bronchitis (Infections and infestations) | 25 | 0
Lower respiratory tract infection (Infections and infestations) | 11 | 2
Oral candidiasis (Infections and infestations) | 15 | 0
Oral herpes (Infections and infestations) | 10 | 2
Pneumonia (Infections and infestations) | 21 | 2
Respiratory tract infection (Infections and infestations) | 9 | 1
Sinusitis (Infections and infestations) | 23 | 3
Upper respiratory tract infection (Infections and infestations) | 47 | 9
Urinary tract infection (Infections and infestations) | 18 | 6
Contusion (Injury, poisoning and procedural complications) | 18 | 3
Infusion related reaction (Injury, poisoning and procedural complications) | 30 | 23
Alanine aminotransferase increased (Investigations) | 19 | 2
Aspartate aminotransferase increased (Investigations) | 14 | 2
Neutrophil count decreased (Investigations) | 16 | 2
Platelet count decreased (Investigations) | 9 | 1
Weight decreased (Investigations) | 28 | 5
Decreased appetite (Metabolism and nutrition disorders) | 37 | 7
Dehydration (Metabolism and nutrition disorders) | 14 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 15 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 32 | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 11 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 12 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 19 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 28 | 11
Muscle spasms (Musculoskeletal and connective tissue disorders) | 18 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 13 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 15 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 19 | 5
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 | 3
Dizziness (Nervous system disorders) | 17 | 5
Dysgeusia (Nervous system disorders) | 11 | 3
Headache (Nervous system disorders) | 37 | 9
Hypoaesthesia (Nervous system disorders) | 10 | 1
Neuropathy peripheral (Nervous system disorders) | 11 | 6
Paraesthesia (Nervous system disorders) | 11 | 4
Peripheral sensory neuropathy (Nervous system disorders) | 6 | 5
Anxiety (Psychiatric disorders) | 15 | 2
Confusional state (Psychiatric disorders) | 10 | 0
Insomnia (Psychiatric disorders) | 30 | 12
Cough (Respiratory, thoracic and mediastinal disorders) | 60 | 18
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 9 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 34 | 11
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9 | 6
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 11 | 6
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 17 | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 17 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 12 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 11 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 17 | 10
Pruritus (Skin and subcutaneous tissue disorders) | 21 | 6
Rash (Skin and subcutaneous tissue disorders) | 36 | 7
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 12 | 0
Hypertension (Vascular disorders) | 21 | 6
Hypotension (Vascular disorders) | 14 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2017-08-30): https://cdn.clinicaltrials.gov/large-docs/21/NCT01659021/Prot_000.pdf
  • Statistical Analysis Plan (2014-09-29): https://cdn.clinicaltrials.gov/large-docs/21/NCT01659021/SAP_001.pdf